CLINICAL TRIAL: NCT03713346
Title: Comparing the Digestion of Milk With Different Beta-casein Protein Content by Dairy Intolerant Persons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Dennis A. Savaiano, Virginia Claypool Meredith Professor of Nutrition Policy, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1710019781
Record Dates: First submitted 2018-04-04; First posted 2018-10-19 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Dairy Intolerance
Keywords: lactose; dairy; intolerance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactose digester (Other)
  Interventions: Other: Lactose free milk; Other: Jersey milk; Other: High A1 β-casein milk; Other: High A2 β-casein milk
- Lactose maldigester (Other)
  Interventions: Other: Lactose free milk; Other: Jersey milk; Other: High A1 β-casein milk; Other: High A2 β-casein milk

INTERVENTIONS:
Other: Lactose free milk — Single dose of lactose free milk
Other: Jersey milk — Single dose of jersey milk
Other: High A1 β-casein milk — Single dose of high A1 β-casein milk (commercial milk)
Other: High A2 β-casein milk — Single dose of A2 β-casein milk

SUMMARY:
Persons with dairy intolerance may experience cramps/abdominal pain, bloating, flatulence, acute diarrhea, or fecal urgency when they ingest excessive amounts of lactose. The intensity of these conditions can be mild or severe and likely depends on numerous variables including dose, transit time, intestinal residual lactase activity and microbiome potential to ferment lactose. Jersey cattle produce milk containing high levels of the A2 β-casein protein . There are claims that high A2 β-casein milk is more easily digested by people who are lactose maldigesters . We propose to conduct a double-blinded, randomized, controlled trial to determine if high A2 β-casein milk from Jersey cattle is actually better digested and tolerated by lactose maldigesters.

DETAILED DESCRIPTION:
Persons with dairy intolerance may experience cramps/abdominal pain, bloating, flatulence, acute diarrhea, or fecal urgency when they ingest excessive amounts of lactose. The intensity of these conditions can be mild or severe and likely depends on numerous variables including dose, transit time, intestinal residual lactase activity and microbiome potential to ferment lactose. Jersey cattle produce milk containing high levels of the A2 β-casein protein . There are claims that high A2 β-casein milk is more easily digested by people who are lactose maldigesters . We propose to conduct a double-blinded, randomized, controlled trial to determine if high A2 β-casein milk from Jersey cattle is actually better digested and tolerated by lactose maldigesters.

This proposed protocol comparing the dairy intolerance symptoms from milks containing predominantly the A1 variant versus A2 variant will establish if high A2 milk is better digested and/or tolerated than high A1 milk.

Participants will be asked to consume four different commercially available milks in random order. The samples will be fed for breakfast separated by at least 10 days, after overnight fasts. The commercial milk treatments will include; high A1 β-casein milk (commercial milk), high A2 β-casein milk, Jersey cattle milk (which contains a mixture of A1 and A2 β-casein), and a lactose free milk control. Milk will be 2% fat content to control for transit. Each subject will be fed milk containing 0.5g lactose per kg body weight. There will be two arms in this study: dairy intolerant who are lactose maldigesters, and dairy intolerant who are lactose digesters.

ELIGIBILITY:
Inclusion Criteria:

1. Ability/desire to provide informed consent
2. Aged 18 to 65 years of age inclusive at screening
3. Current or recent history of intolerance to and avoidance of milk of at least one month duration (by self-report and self-reported symptoms).
4. Agrees to refrain from all other treatments and products used for lactose intolerance (e.g., Lactaid® Dietary Supplements) during study involvement
5. Willing to return for all study visits and complete all study related procedures, including fasting before and during the hydrogen breath tests
6. Qualifying Lactose Challenge Symptom Score:

(4 symptom categories with severity measured on from 0 to 5) as defined by one of the following:

1. At least one score of "moderately severe" or "severe" on a single symptom during the 6 hour HBT test;
2. A score of "moderate" or greater for a single symptom on at least two (2) time points during the 6 hour HBT test;
3. At least one "moderate" score or greater on each of two symptoms during the 6 hour HBT test 7. Hydrogen concentration of at least 20 parts per million greater than baseline at least 2 time points during the screening hydrogren breath test 8. Able to understand and provide written informed consent in English

Exclusion Criteria:

1. Allergic to milk
2. Currently pregnant
3. Currently lactating
4. Cigarette smoking or other use of tobacco or nicotine containing products within 3 months of screening
5. Diagnosed with any of the following disorders known to be associated with abnormal gastrointestinal motility such as; Gastroparesis, amyloidosis, neuromuscular diseases (including Parkinson's disease), collagen vascular diseases, alcoholism, uremia, malnutrition, or untreated hypothyroidism
6. History of surgery that alters the normal function of the gastrointestinal tract including, but not limited to: gastrointestinal bypass surgery, bariatric surgery, gastric banding, vagotomy, fundoplication, pyloroplasty [Note: history of uncomplicated abdominal surgeries such as removal of an appendix more than 12 months prior to screening will not be excluded]
7. Past or present : Organ transplant, chronic pancreatitis, pancreatic insufficiency, symptomatic biliary disease, Celiac disease, chronic constipation, diverticulosis, inflammatory bowel disease (IBD), ulcerative colitis (UC), Crohn's disease (CD), small intestine bacterial overgrowth syndrome (SIBO), gastroparesis, gastro-esophageal reflux disease (GERD), Irritable Bowel Syndrome (IBS) or any other medical condition with symptoms that could confound collection of adverse events.
8. Active ulcers, or history of severe ulcers
9. Diabetes mellitus (type 1 and type 2)
10. Congestive Heart Failure (CHF)
11. Human Immunodeficiency Virus (HIV), Hepatitis B or Hepatitis C
12. BMI > 35 kg/m2
13. Recent bowel preparation for endoscopic or radiologic investigation within four weeks of screening (e.g., colonoscopy prep)
14. Use of concurrent therapy(ies) or other products (e.g., laxatives, stool softeners, Pepto Bismol®, Lactaid® Dietary Supplements) used for symptoms of lactose intolerance within 7 days of screening
15. Chronic antacid and/or PPI use
16. Recent use of systemic antibiotics defined as use within 30 days prior to screening
17. Recent high colonic enema, defined as use within 30 days prior to screening
18. Any concurrent disease or symptoms which may interfere with the assessment of the cardinal symptoms of lactose intolerance (i.e., gas, diarrhea, bloating, cramps, stomach pain)
19. History of ethanol (alcohol) and/or drug abuse in the past 12 months
20. Currently undergoing chemotherapy
21. Use of any investigational drug or participation in any investigational study within 30 days prior to screening
22. Prior enrollment in this study
23. Any other conditions/issues noted by the study staff and/or Principal Investigator that would impact participation and/or protocol compliance

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Differences in AUC ΔH2 concentrations | Within the 6 hours following the milk challenge
  Differences in AUC ΔH2 concentrations (primary outcomes) among milk phases is examined by repeated-measures analysis of variance (ANOVA)

SECONDARY OUTCOMES:
Differences within each of the symptom categories | Within the 6 hours following the milk challenge
  Repeated-measures ANOVA is also used to test for differences within each of the symptom categories (secondary outcomes) after transforming to correct for nonstationary variance. For both the H2 concentrations and symptom levels, to be able to detect differences between every single treatment, pairwise differences are examined using least significant difference (LSD).

CONTACTS AND LOCATIONS:
Overall Officials: Dennis A Savaiano, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Background] Briet F, Pochart P, Marteau P, Flourie B, Arrigoni E, Rambaud JC. Improved clinical tolerance to chronic lactose ingestion in subjects with lactose intolerance: a placebo effect? Gut. 1997 Nov;41(5):632-5. doi: 10.1136/gut.41.5.632. PMID 9414969
- [Background] Dairy Farmer. (2011). Specialist A2 milk venture. Cengage Learning, Inc. 2.
- [Background] Brown-Esters, O., Mc Namara, P., & Savaiano, D. (2012). Dietary and biological factors influencing lactose intolerance. International Dairy Journal, 22(2), 98-103.
- [Background] Davies, D.T. & Law, A.J.R. (1980). The content and composition of creamery milks in south-west Scotland. J Dairy Res, 47, 80-90.
- [Background] Carroccio A, Montalto G, Cavera G, Notarbatolo A. Lactose intolerance and self-reported milk intolerance: relationship with lactose maldigestion and nutrient intake. Lactase Deficiency Study Group. J Am Coll Nutr. 1998 Dec;17(6):631-6. doi: 10.1080/07315724.1998.10718813. PMID 9853544
- [Background] de Silva P, Rachman S. Human food aversions: nature and acquisition. Behav Res Ther. 1987;25(6):457-68. doi: 10.1016/0005-7967(87)90053-2. No abstract available. PMID 3426508
- [Background] Dehkordi N, Rao DR, Warren AP, Chawan CB. Lactose malabsorption as influenced by chocolate milk, skim milk, sucrose, whole milk, and lactic cultures. J Am Diet Assoc. 1995 Apr;95(4):484-6. doi: 10.1016/S0002-8223(95)00126-3. No abstract available. PMID 7699193
- [Background] DOELL RG, KRETCHMER N. Studies of small intestine during development. I. Distribution and activity of beta-galactosidase. Biochim Biophys Acta. 1962 Aug 13;62:353-62. doi: 10.1016/0006-3002(62)90097-5. No abstract available. PMID 13886893
- [Background] Gilliland SE, Kim HS. Effect of viable starter culture bacteria in yogurt on lactose utilization in humans. J Dairy Sci. 1984 Jan;67(1):1-6. doi: 10.3168/jds.S0022-0302(84)81260-6. PMID 6707296
- [Background] Gustavsson F, Buitenhuis AJ, Johansson M, Bertelsen HP, Glantz M, Poulsen NA, Lindmark Mansson H, Stalhammar H, Larsen LB, Bendixen C, Paulsson M, Andren A. Effects of breed and casein genetic variants on protein profile in milk from Swedish Red, Danish Holstein, and Danish Jersey cows. J Dairy Sci. 2014;97(6):3866-77. doi: 10.3168/jds.2013-7312. Epub 2014 Apr 3. PMID 24704225
- [Background] Haverberg L, Kwon PH, Scrimshaw NS. Comparative tolerance of adolescents of differing ethic backgrounds to lactose-containing and lactose-free dairy drinks. I. Initial experience with a double-blind procedure. Am J Clin Nutr. 1980 Jan;33(1):17-21. doi: 10.1093/ajcn/33.1.17. PMID 7188826
- [Background] Hayes, J. (2014). Farm Weekly. A2 milk drinkers may get less gut aches. Global Reference on the Environment, Energy, and Natural Resources.
- [Background] He T, Priebe MG, Harmsen HJ, Stellaard F, Sun X, Welling GW, Vonk RJ. Colonic fermentation may play a role in lactose intolerance in humans. J Nutr. 2006 Jan;136(1):58-63. doi: 10.1093/jn/136.1.58. PMID 16365059
- [Background] Hertzler SR, Savaiano DA. Colonic adaptation to daily lactose feeding in lactose maldigesters reduces lactose intolerance. Am J Clin Nutr. 1996 Aug;64(2):232-6. doi: 10.1093/ajcn/64.2.232. PMID 8694025
- [Background] Ho S, Woodford K, Kukuljan S, Pal S. Comparative effects of A1 versus A2 beta-casein on gastrointestinal measures: a blinded randomised cross-over pilot study. Eur J Clin Nutr. 2014 Sep;68(9):994-1000. doi: 10.1038/ejcn.2014.127. Epub 2014 Jul 2. PMID 24986816
- [Background] Johnson AO, Semenya JG, Buchowski MS, Enwonwu CO, Scrimshaw NS. Correlation of lactose maldigestion, lactose intolerance, and milk intolerance. Am J Clin Nutr. 1993 Mar;57(3):399-401. doi: 10.1093/ajcn/57.3.399. PMID 8438774
- [Background] Johnson AO, Semenya JG, Buchowski MS, Enwonwu CO, Scrimshaw NS. Adaptation of lactose maldigesters to continued milk intakes. Am J Clin Nutr. 1993 Dec;58(6):879-81. doi: 10.1093/ajcn/58.6.879. PMID 8249871
- [Background] Kolars JC, Levitt MD, Aouji M, Savaiano DA. Yogurt--an autodigesting source of lactose. N Engl J Med. 1984 Jan 5;310(1):1-3. doi: 10.1056/NEJM198401053100101. PMID 6417539
- [Background] Kretchmer N. On the homology between human development and pediatrics. Pediatr Res. 1968 Jul;2(4):283-6. doi: 10.1203/00006450-196807000-00007. No abstract available. PMID 5669665
- [Background] Kretchmer N. Lactose and lactase--a historical perspective. Gastroenterology. 1971 Dec;61(6):805-13. No abstract available. PMID 4947662
- [Background] Lee CM, Hardy CM. Cocoa feeding and human lactose intolerance. Am J Clin Nutr. 1989 May;49(5):840-4. doi: 10.1093/ajcn/49.5.840. PMID 2718917
- [Background] Leichter J. Comparison of whole milk and skim milk with aqueous lactose solution in lactose tolerance testing. Am J Clin Nutr. 1973 Apr;26(4):393-6. doi: 10.1093/ajcn/26.4.393. No abstract available. PMID 4740264
- [Background] Lerebours E, N'Djitoyap Ndam C, Lavoine A, Hellot MF, Antoine JM, Colin R. Yogurt and fermented-then-pasteurized milk: effects of short-term and long-term ingestion on lactose absorption and mucosal lactase activity in lactase-deficient subjects. Am J Clin Nutr. 1989 May;49(5):823-7. doi: 10.1093/ajcn/49.5.823. PMID 2497632
- [Background] Logue AW, Ophir I, Strauss KE. The acquisition of taste aversions in humans. Behav Res Ther. 1981;19(4):319-33. doi: 10.1016/0005-7967(81)90053-x. No abstract available. PMID 7271698
- [Background] Martini MC, Savaiano DA. Reduced intolerance symptoms from lactose consumed during a meal. Am J Clin Nutr. 1988 Jan;47(1):57-60. doi: 10.1093/ajcn/47.1.57. PMID 3122554
- [Background] Moore BJ. Dairy Foods: Are They Politically Correct? Nutr Today. 2003 May-Jun;38(3):82-90. PMID 12813186
- [Background] Newcomer AD, McGill DB, Thomas PJ, Hofmann AF. Tolerance to lactose among lactase-deficient American Indians. Gastroenterology. 1978 Jan;74(1):44-6. PMID 336450
- [Background] Ng-Kwai-Hang KF & Grosclaude F. (2003). Genetic polymorphism of milk proteins. Advanced Dairy Chemistry, 1, 739-816.
- [Background] Perets, T., Shporn, E., Bareli, Y., Kelner, Y., Levy, S., Aizic, S., Pakanaev, L., Niv, Y., & Dickman, R. (2013). Clinical Accuracy and Usefulness of the Lactose Intolerance Quick Test for the Diagnosis of Lactose Malabsorption. Gastroenterology, 144(5), S473
- [Background] Rask Pedersen E, Jensen BH, Jensen HJ, Keldsbo IL, Hylander Moller E, Norby Rasmussen S. Lactose malabsorption and tolerance of lactose-hydrolyzed milk. A double-blind controlled crossover study. Scand J Gastroenterol. 1982 Oct;17(7):861-4. doi: 10.3109/00365528209181106. PMID 6818684
- [Background] Reasoner J, Maculan TP, Rand AG, Thayer WR Jr. Clinical studies with low-lactose milk. Am J Clin Nutr. 1981 Jan;34(1):54-60. doi: 10.1093/ajcn/34.1.54. PMID 6893787
- [Background] Rosensweig NS. Adult human milk intolerance and intestinal lactase deficiency. A review. J Dairy Sci. 1969 May;52(5):585-7. doi: 10.3168/jds.S0022-0302(69)86611-7. No abstract available. PMID 4902392
- [Background] Savaiano DA, Levitt MD. Milk intolerance and microbe-containing dairy foods. J Dairy Sci. 1987 Feb;70(2):397-406. doi: 10.3168/jds.S0022-0302(87)80023-1. PMID 3553256
- [Background] Savaiano, D., Hertzler, S., Jackson, A. J., & Suarez, F. L. (2001). Nutrient considerations in lactose intolerance. In A. M. Coulston, C. L. Rock, & E. R. Monsen (Eds.), Nutrition in the prevention and treatment of disease San Diego, CA, USA: Academic Press. 563-575
- [Background] Savaiano DA, AbouElAnouar A, Smith DE, Levitt MD. Lactose malabsorption from yogurt, pasteurized yogurt, sweet acidophilus milk, and cultured milk in lactase-deficient individuals. Am J Clin Nutr. 1984 Dec;40(6):1219-23. doi: 10.1093/ajcn/40.6.1219. PMID 6439026
- [Background] Scrimshaw NS, Murray E. [Lactose tolerance and milk consumption: myths and realities]. Arch Latinoam Nutr. 1988 Sep;38(3):543-67. Spanish. PMID 3155250
- [Background] Shermak MA, Saavedra JM, Jackson TL, Huang SS, Bayless TM, Perman JA. Effect of yogurt on symptoms and kinetics of hydrogen production in lactose-malabsorbing children. Am J Clin Nutr. 1995 Nov;62(5):1003-6. doi: 10.1093/ajcn/62.5.1003. PMID 7572723
- [Background] Simoons FJ. The geographic hypothesis and lactose malabsorption. A weighing of the evidence. Am J Dig Dis. 1978 Nov;23(11):963-80. doi: 10.1007/BF01263095. PMID 362904
- [Background] Solomons NW, Guerrero AM, Torun B. Dietary manipulation of postprandial colonic lactose fermentation: II. Addition of exogenous, microbial beta-galactosidases at mealtime. Am J Clin Nutr. 1985 Feb;41(2):209-21. doi: 10.1093/ajcn/41.2.209. PMID 3918430
- [Background] Suarez FL, Adshead J, Furne JK, Levitt MD. Lactose maldigestion is not an impediment to the intake of 1500 mg calcium daily as dairy products. Am J Clin Nutr. 1998 Nov;68(5):1118-22. doi: 10.1093/ajcn/68.5.1118. PMID 9808231
- [Background] Suarez FL, Savaiano DA, Levitt MD. Review article: the treatment of lactose intolerance. Aliment Pharmacol Ther. 1995 Dec;9(6):589-97. doi: 10.1111/j.1365-2036.1995.tb00427.x. PMID 8824645
- [Background] Suarez FL, Savaiano D, Arbisi P, Levitt MD. Tolerance to the daily ingestion of two cups of milk by individuals claiming lactose intolerance. Am J Clin Nutr. 1997 May;65(5):1502-6. doi: 10.1093/ajcn/65.5.1502. PMID 9129483
- [Background] Suchy FJ, Brannon PM, Carpenter TO, Fernandez JR, Gilsanz V, Gould JB, Hall K, Hui SL, Lupton J, Mennella J, Miller NJ, Osganian SK, Sellmeyer DE, Wolf MA. National Institutes of Health Consensus Development Conference: lactose intolerance and health. Ann Intern Med. 2010 Jun 15;152(12):792-6. doi: 10.7326/0003-4819-152-12-201006150-00248. Epub 2010 Apr 19. No abstract available. PMID 20404261
- [Background] Swagerty DL Jr, Walling AD, Klein RM. Lactose intolerance. Am Fam Physician. 2002 May 1;65(9):1845-50. PMID 12018807
- [Background] Truswell AS. The A2 milk case: a critical review. Eur J Clin Nutr. 2005 May;59(5):623-31. doi: 10.1038/sj.ejcn.1602104. PMID 15867940
- [Background] Welsh JD, Hall WH. Gastric emptying of lactose and milk in subjects with lactose malabsorption. Am J Dig Dis. 1977 Dec;22(12):1060-3. doi: 10.1007/BF01072857. PMID 579279